CLINICAL TRIAL: NCT07180056
Title: Efficacy and Safety of Adjuvant CDK4/6 Inhibitors in Patients With Hormone Receptor-positive/Human Epidermal Growth Factor Receptor 2-negative Breast Cancer: a Real-world Study
Brief Title: Adjuvant CDK4/6 Inhibitor Use in HR+/HER2- Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Wenjin Yin (Other)
Responsible Party: Sponsor-Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: LY2025-108-B
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adjuvant CDK4/6 inhibitor: CDK4/6 inhibitors are drugs that block cell division in cancer cells. They are used with hormonal therapy for hormone receptor-positive breast cancer and may improve survival.
  Interventions: Drug: CDK4/6 inhibitor

INTERVENTIONS:
Drug: CDK4/6 inhibitor — abemaciclib OR ribociclib

SUMMARY:
To evaluate the efficacy and safety of adjuvant CDK4/6 inhibitors in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and older
* Patients with pathologically confirmed breast cancer without distant metastasis or local recurrence
* HR+/HER2-
* ECOG 0-3
* Subjects meeting current guideline recommendations and planning to receive adjuvant CDK4/6 inhibitors

Exclusion Criteria:

* During pregnancy or lactation
* Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients meeting current guideline recommendations and planning to receive adjuvant CDK4/6 inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 229 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (iDFS) | From the date of surgery until time of event up to 2 years.
  Invasive disease-free survival time is defined as the time from date of randomization until the first invasive disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, distant recurrence and death from any cause.

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | From the date of surgery until time of event up to 2 years
  Disease-free survival time is defined as the time from date of surgery until the first disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, non-breast primary invasive cancer, ductal carcinoma in situ (DCIS),or distant recurrence and death from any cause.
Overall Survival (OS) | From the date of surgery until time of event up to 2 years
  Overall survival is defined as the time from surgery to death from any cause.
Adverse events | From the date of starting CDK4/6 inhibitor to the end of the treatment (up to approximately 3 years)
  Adverse events will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital,School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No